CLINICAL TRIAL: NCT00793858
Title: A Pilot Investigation of the Nasal Mucosal Absorption, Retention, and Metabolism of Ciclesonide When Administered as a Hypotonic Versus an Isotonic Formulation of Ciclesonide Nasal Spray When Each Formulation Is Administered to Currently Symptomatic Patients (18 Years or Older) With Documented Perennial Allergic Rhinitis (PAR).
Brief Title: A Pilot Investigation of Ciclesonide When Administered as a Hypotonic Versus an Isotonic Formulation of Ciclesonide Nasal Spray
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Cost prohibitive and company withdrew support.
Sponsor: University of Chicago (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 16651A (SEP 1)
Record Dates: First submitted 2008-11-14; First posted 2008-11-19 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Active Comparator): placebo in left nostril, isotonic ciclesonide in right
  Interventions: Drug: placebo, isotonic ciclesonide, hypotonic ciclesonide
- 2 (Active Comparator): hypotonic ciclesonide in left nostril, placebo in right
  Interventions: Drug: placebo, isotonic ciclesonide, hypotonic ciclesonide
- 3 (Active Comparator): hypotonic ciclesonide in right and left nostrils
  Interventions: Drug: placebo, isotonic ciclesonide, hypotonic ciclesonide
- 4 (Active Comparator): isotonic ciclesonide in both right and left nostrils
  Interventions: Drug: placebo, isotonic ciclesonide, hypotonic ciclesonide
- 6 (Placebo Comparator): placebo in both right and left nostrils
  Interventions: Drug: placebo, isotonic ciclesonide, hypotonic ciclesonide
- 5 (Active Comparator): isotonic ciclesonide in left nostril and hypotonic ciclesonide in right
  Interventions: Drug: placebo, isotonic ciclesonide, hypotonic ciclesonide

INTERVENTIONS:
Drug: placebo, isotonic ciclesonide, hypotonic ciclesonide — 200mcg/nostril

SUMMARY:
The purpose of this study is to measure the amount of a nasal steroid spray (ciclesonide) absorbed by the tissue in the nose 2 hours after having this study drug sprayed in the nose

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age or older.
2. History of perennial allergic rhinitis for at least 1 year prior to screening.
3. Positive skin test to perennial allergen.

Exclusion Criteria:

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Upper respiratory infection within 14 days of study start.
4. Active asthma requiring treatment with inhaled or systemic steroids.
5. Use of any form of nasal spray during the previous month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
levels of ciclesonide in biopsy tissue | 2 hours post study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States